CLINICAL TRIAL: NCT05737095
Title: Study of the Feasibility of Early Lung Ultrasound in Neonatal Respiratory Distress in Premature Newborns Born Between 32 Weeks of Amenorrhea and 36 Weeks Plus 6 Days of Amenorrhea, Hospitalized in the Neonatal Pediatrics and Intensive Care Units of the Dijon University Hospital
Acronym: REchoPP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: TERNOY-LANZINI 2022
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Neonatal Respiratory Distress; Preterm Birth
MeSH Terms: conditions — Pulmonary Atelectasis; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Premature infants: premature infants born between 32 and 36 weeks of amenorrhea + 6 days hospitalized for respiratory distress
  Interventions: Procedure: Pulmonary ultrasound

INTERVENTIONS:
Procedure: Pulmonary ultrasound — Within 6 hours of admission to Neonatal Pediatrics and Intensive Care

SUMMARY:
Monocentric study carried out in the Neonatal and Intensive Care Units of the Dijon University Hospital.

The objective is to evaluate the feasibility of performing a pulmonary ultrasound within 6 hours after admission in premature infants born between 32 weeks of amenorrhea and 36 weeks of amenorrhea + 6 days who are hospitalized for initial respiratory distress.

Pulmonary ultrasound is performed within 6 hours of admission and an ultrasound score is calculated according to the images observed.

Continued management according to protocols without taking into account the ultrasound data.

Follow-up of patients until discharge from hospital or D28 of life (whichever comes first)

ELIGIBILITY:
Inclusion Criteria:

* Verbal consent from at least one legal guardian
* Premature infant (between 32 weeks of amenorrhea and 36 weeks of amenorrhea + 6 days) admitted for neonatal respiratory distress that began in the first 2 hours of life
* Hospitalized at the Dijon University Hospital in the Neonatal Pediatrics and Intensive Care Units

Exclusion Criteria:

* individual is not affiliated to the national health care system
* major intrathoracic or abdominal malformation

Ages: 0 Hours to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-11-27 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Number of infants receiving a lung ultrasound within 6 hours of admission divided by the number of infants meeting the inclusion criteria | Within 6 hours of admission
  Number of infants receiving a lung ultrasound within 6 hours of admission divided by the number of infants meeting the inclusion criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No